## Ethical board/consent

(S2)

## Informed consent for participation in a health care research project

Project's title: The effect of a heel-unloading orthosis in short-term treatment of calcaneus fractures on physical function, quality of life and return to work – a randomized controlled trial

## **Declaration by the participant/patient:**

I have received written and oral information and I know enough about the purpose, method, advantages and disadvantages to say yes to participate.

I know it's voluntary to participate and that I can always withdraw my consent without losing my current or future rights to treatment.

I agree to participate in the research project and have received a copy of this consent sheet as well as a copy of the written information about the project for its own use.

| Participant's name: | |
|---|---|
| Date: | Signature: |
| informed. Would you lik | information comes forward about you in the research project, you will be to disclose information about new essential health information that appears in ease select here:(set x) |
| Do you want to be infor | med about the results of the research project and any consequences for you?: |
| Yes(set x) | No(set x) |
| Declaration of the person providing information: | |
| I declare that the subject | ct has received oral and written information about the trial. |
| In my conviction, sufficient information has been provided for a decision to participate in the trial. The name of the person providing information: | |
| Date: | Signature: |
| Project identification: (i | .e. EB project-ID, EudraCT nr., version nr./date or similar) 61555 |

Standard form Informed consent prepared by the Ethical board of the Region of Southern Denmark, August 2016.